CLINICAL TRIAL: NCT02322606
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of TAK-137 in Healthy Subjects
Brief Title: A Phase 1, Single and Multiple Dose Study of TAK-137
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-137/CPH-001; U1111-1162-5936 (Registry Identifier: WHO)
Record Dates: First submitted 2014-10-28; First posted 2014-12-23 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Japanese Adult Male
MeSH Terms: interventions — TAK-137; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1: TAK-137 5 mg, TAK-137 placebo (Other): Single-dose administration in a fasting state
  Interventions: Drug: TAK-137 5 mg tablet, TAK-137 placebo tablet
- Cohort 2: TAK-137 10 mg, TAK-137 placebo tablet (Other): Single-dose administration in a fasting state
  Interventions: Drug: TAK-137 5 mg tablet, TAK-137 placebo tablet
- Cohort 3: TAK-137 20 mg or TAK-137 2 mg + TAK-137 placebo (Other): Single-dose administration in a fasting state
  Interventions: Drug: TAK-137 5 mg tablet, TAK-137 placebo tablet or TAK-137 0.5 mg tablet, TAK-137 placebo tablet
- Cohort 4: TAK-137 5mg, TAK-137 placebo (Other): Once daily for 7 days in a fasting state
  Interventions: Drug: TAK-137 5mg tablet, TAK-137 placebo tablet
- Cohort 5: TAK-137 10 mg, TAK-137 placebo (Other): Once daily for 7 days in a fasting state
  Interventions: Drug: TAK-137 5 mg tablet, TAK-137 placebo tablet
- Cohort 6: TAK-137 15 mg, TAK-137 placebo (Other): Once daily for 7 days in a fasting state
  Interventions: Drug: TAK-137 5mg tablet, TAK-137 placebo tablet

INTERVENTIONS:
Drug: TAK-137 5 mg tablet, TAK-137 placebo tablet
  Arms: Cohort 1: TAK-137 5 mg, TAK-137 placebo
Drug: TAK-137 5 mg tablet, TAK-137 placebo tablet
  Arms: Cohort 2: TAK-137 10 mg, TAK-137 placebo tablet
Drug: TAK-137 5 mg tablet, TAK-137 placebo tablet or TAK-137 0.5 mg tablet, TAK-137 placebo tablet
  Arms: Cohort 3: TAK-137 20 mg or TAK-137 2 mg + TAK-137 placebo
Drug: TAK-137 5mg tablet, TAK-137 placebo tablet
  Arms: Cohort 4: TAK-137 5mg, TAK-137 placebo
Drug: TAK-137 5 mg tablet, TAK-137 placebo tablet
  Arms: Cohort 5: TAK-137 10 mg, TAK-137 placebo
Drug: TAK-137 5mg tablet, TAK-137 placebo tablet
  Arms: Cohort 6: TAK-137 15 mg, TAK-137 placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of TAK-137 in healthy male subjects.

DETAILED DESCRIPTION:
This study is a phase 1, randomized, placebo-controlled, double-blind, multiple ascending dose study in Japanese healthy male participants to assess the safety, tolerability and PK following single and multiple oral doses of TAK-137.

This study is composed of 2 parts, a Single Dose part (Cohorts 1 to 3) and a Multiple Dose part (Cohorts 4 to 6). Up to 48 participants will be enrolled.

Single dose part (Cohorts 1-3): Single Dose, 3 dose levels, Placebo-Controlled, Randomized, Double-Blind.

Each cohort will include 8 participants. Participants will be randomly assigned to either TAK-137 or placebo treatment group within each cohort with an allocation ratio of 6:2.

The planned dose levels to be studied are 5, 10 and 20 mg. The principal investigator will consult with the sponsor and the medical specialist as needed and will determine go/no-go for the next cohort.. The dose in Cohorts 3 may be reduced to 2 mg/day instead of 20 mg/day if the principal investigator, in consultation with the sponsor, considers it appropriate.

Multiple dose Part (Cohorts 4-6): Multiple Dose, 3 dose levels, Placebo-Controlled, Randomized, Double-Blind.

Each cohort will include 8 participants. Participants will be randomly assigned to either TAK-137 or placebo treatment group within each cohort with an allocation ratio of 6:2.

The planned dose levels to be studied are 5, 10,and 15 mg, however for Cohort 5 and 6, the dose level may be amended based on the safety and tolerability data obtained from either Cohorts 1-4 from this study or emerging data from the multiple rising dose study conducted, in parallel in the United Sates (TAK-137_102). The principle investigator, in consultation with the sponsor, will determine the dose levels for cohorts 5 and 6 (Not exceeding 20mg).

ELIGIBILITY:
Inclusion Criteria:

* Participant eligibility is determined according to the following criteria prior to entry into the study:

  * In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
  * The participant signs and dates a written, ICF and any required privacy authorization prior to the initiation of any study procedures.
  * The participant is a healthy Japanese adult male volunteer.
  * The participant is between 20 and 45 years of age at the time of informed consent.
  * The participant has a body weight of at least 50 kg and has a body mass index (BMI) between 18.5 and 24.9 kg/m2 at the time of screening and baseline (Day -1).
  * A male participant who is sexually active with a female partner of childbearing potential agrees to use adequate contraception after signing the ICF for up to 12 weeks from the last dose.

Exclusion Criteria:

* Any participant who meets any of the following criteria will not qualify for entry into the study:

  * The participant has received any investigational drugs within 30 days prior to the first study drug administration.
  * The participant has received TAK-137 in a previous clinical study.
  * The participant is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
  * The participant has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic or endocrine disease or other abnormality which may impact the ability of the participant to participate or potentially confound the study results.
  * The participant has previously had a seizure or convulsion (lifetime), including absence seizure and febrile convulsion
  * The participant has a history of psychiatric disorders.
  * The participant has a known hypersensitivity to medication(s) or food(s).
  * The participant has positive results in the urine drug screening test at screening.
  * The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 2 years prior to the screening or is unwilling to agree to abstain from alcohol and drugs throughout the study period.
  * The participant has taken any excluded medication, supplements, or food products listed in the Excluded Medications and Dietary Products during the screening period, or requires such medication or food during the study.
  * The participant intends to donate sperm from the signing of ICF to 12 weeks after the last dose.
  * The participant has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (i.e., a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn, or any surgical intervention, [e.g. gastrectomy, cholecystectomy, etc.]).
  * The subject has a history of cancer.
  * The subject has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody/antigen, or serological reactions for syphilis at screening.
  * The subject has poor peripheral venous access.
  * The subject has undergone whole blood collection of at least 200 mL within 4 weeks (28 days) or at least 400 mL within 12 weeks (84 days) prior to the first study drug administration.
  * The participant has undergone whole blood collection of at least 800 mL in total within 52 weeks (364 days) prior to the first study drug administration.
  * The participant has undergone blood component collection within 2 weeks (14 days) prior to the first study drug administration.
  * The participant has any clinically significant ECG abnormality at time of screening or baseline (Day -1).
  * The participant has abnormal screening or baseline (Day -1) laboratory values that suggest a clinically significant underlying disease, or the participant has the following lab abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 × the upper limits of normal (ULN).
  * The participant has an abnormal EEG during screening
  * The participant is at risk for suicide based on the investigator's determination.
  * The participant who, in the opinion of the investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Frequencies of Adverse events (Single dose Part) | Up to 8 days
  The frequencies of all adverse events observed during the observation period will be tabulated by type and seriousness, and causal relationship to TAK-137. Adverse events are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product, reported from the first dose to the last dose of TAK-137.
Frequencies of Adverse events (Multiple dose Part) | Up to 14 days
  The frequencies of all adverse events observed during the observation period will be tabulated by type and seriousness, and causal relationship to TAK-137. Adverse events are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product, reported from the first dose to the last dose of TAK-137.
Descriptive statistics (mean, SD, median, minimum and maximum) of changes from baseline for vital sign measurements at least once post-dose (Single dose Part) | Up to 8 days
Descriptive statistics (mean, SD, median, minimum and maximum) of changes from baseline for vital sign measurements at least once post-dose (Multiple dose Part) | Up to 9 days
Descriptive statistics (mean, SD, median, minimum and maximum) of changes from baseline for body weight measurements at least once post-dose (Single dose Part) | Up to 8 days
Descriptive statistics (mean, SD, median, minimum and maximum) of changes from baseline for body weight measurements at least once post-dose (Multiple dose Part) | Up to 9 days
Percentage of participants with abnormal and clinically significant judged by investigator for electrocardiogram measurements at least once post-dose (Single dose Part) | Up to 8 days
  The percentage of participants with abnormal and clinically significant judged by investigator, electrocardiogram measurements during the study period.
Percentage of participants with abnormal and clinically significant judged by investigator for electrocardiogram measurements at least once post-dose (Multiple dose Part) | Up to 9 days
  The percentage of participants with abnormal and clinically significant judged by investigator, electrocardiogram measurements during the study period.
Percentage of participants with significantly abnormal (epileptiform) judged by investigator for electroencephalogram measurements at least once post-dose (Single dose Part) | Up to 1 day
  The percentage of participants with significantly abnormal (epileptiform) judged by investigator, electroencephalogram measurements during the study period.
Percentage of participants with significantly abnormal (epileptiform) judged by investigator for electroencephalogram measurements at least once post-dose (Multiple dose Part) | Up to 7 days
  The percentage of participants with significantly abnormal (epileptiform) judged by investigator, electroencephalogram measurements during the study period.
Percentage of participants who meet the markedly abnormal criteria for safety laboratory tests at least once post-dose (Single dose Part) | Up to 8 days
  The percentage of participants with any markedly abnormal, standard safety laboratory values, including hematology and serum chemistries during the study period.
Percentage of participants who meet the markedly abnormal criteria for safety laboratory tests at least once post-dose (Multiple dose Part) | Up to 9 days
  The percentage of participants with any markedly abnorma, standard safety laboratory values, including hematology and serum chemistries during the study period.
Descriptive statistics (mean, SD, median, minimum and maximum) of observed value for Stimulant relapse risk scale (excerpt) (Single dose Part) | Up to 8 days
Descriptive statistics (mean, SD, median, minimum and maximum) of observed value for Stimulant relapse risk scale (excerpt) (Multiple dose Part ) | Up to 9 days

SECONDARY OUTCOMES:
Descriptive statistics (mean, SD, median, minimum and maximum) of pharmacokinetic parameters (AUC(0-168), AUC(0-tlqc), Cmax, Tmax, AUC(0-inf), T1/2, CL/F, Vz/F and MR) for unchanged TAK-137 and its metabolite M-I in plasma (Single dose Part) | Days 1-8
  The pharmacokinetic parameters (AUC(0-168), AUC(0-tlqc), Cmax, Tmax, AUC(0-inf), T1/2, CL/F, Vz/F and MR) will be estimated from a Non-compartmental analysis.
Descriptive statistics (mean, SD, median, min. and max.) of pharmacokinetic parameters for unchanged TAK-137 and its metabolite M-I in plasma (Multiple dose Part) | Days 1-9
  The pharmacokinetic parameters (AUC(0-24), AUC(0-tlqc), Cmax, Tmax, AUC(0-inf), T1/2, CL/F, Vz/F, MR, Cavg, R(AUC), R(Cmax), AI(AUC) and AI(T1/2)) will be estimated from a Non-compartmental analysis.
Descriptive statistics (mean, SD, median, minimum and maximum) of pharmacokinetic parameters (Fe and CLr) for unchanged TAK-137 and its metabolite M-I in urine (Single dose Part) | Days 1-4 (Prior to administration and 0-24, 24-48, 48-72 hours after administration)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Takeda
Locations (1):
- Kagoshima, Kagoshima-ken, Japan